CLINICAL TRIAL: NCT04505241
Title: Evaluating Mechanisms of Action of Adaptive Goal-Setting for Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Evan Forman, Professor of Psychology, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRX-7861
Record Dates: First submitted 2020-08-02; First posted 2020-08-10 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Motivation; Physical Activity Promotion; Behavior Change; Mobile Health
Keywords: Physical Activity; Goal-Setting; Adaptive Interventions; Health-Related Behavior Change
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Half of participants will be randomized to receive text message-delivered adaptive goal-setting (goals change each day) for 6 weeks, and half will receive static goal-setting (goals are fixed) for 6 weeks.
Who Masked: Participant, Investigator
Masking Description: Participants will not be informed of their assigned condition, though may infer it through the types of texts that they receive.
  The principal investigator and outcomes assessor will each be blinded to a participant's assignment while the participant is enrolled in the study, and will be unblinded at the conclusion of the study prior to performing statistical analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive Goal-Setting (Experimental): Participants in this condition will receive daily step goals calculated as the 60th percentile of their last 9 days of available daily steps data. Goals will be transmitted over text message, and will be accompanied by information about the participant's steps on the previous day and whether they met their goal the previous day.
  Interventions: Behavioral: Remotely-delivered physical activity promotion
- Static Goal-Setting (Experimental): Participants in this condition will receive daily a uniform daily goal of 10,000 steps per day. Participants will receive daily texts including information about the participant's steps on the previous day, whether they met their goal the previous day, and encouraging them to continue striving for 10,000 steps each day.
  Interventions: Behavioral: Remotely-delivered physical activity promotion

INTERVENTIONS:
Behavioral: Remotely-delivered physical activity promotion — Over video-call, participants will receive educational content on safely increasing their levels of physical activity (e.g., selecting an appropriate form of exercise, minimizing health risks, the importance of planning), will receive daily text messages (see arm descriptions) for six weeks and complete a 10-15 minute check-in call at the 3-week point of the intervention to assess compliance with daily step goals as well as to help problem-solve barriers to compliance.

SUMMARY:
Behavior modification programs hold promise for increasing levels of physical activity (PA) for individuals who are insufficiently active. However, existing interventions, which typically prescribe uniform PA goals across participants, are limited by their insensitivity to changing individual needs and circumstances over time. An alternative approach is to continuously adjust goal difficulty to match fluctuations in individual performance, or adaptive goal-setting (AGS), which evidence suggests may more effective for increasing PA than non-adaptive approaches. Still, no prior studies have examined the psychological mechanisms targeted by AGS, which limits the ability to further refine and disseminate this technique. In this exploratory study, several candidate mechanisms of AGS (expectancy beliefs about goals, perceived value of goals, affective appraisal of goals, implicit attitudes towards exercise) will be examined. Adult participants interested in increasing their level of physical activity (N = 36) will be randomized to receive 6 weeks of either adaptive goal-setting (AGS) or non-adaptive, static goal-setting (SGS) as part of a remote, low-intensity PA intervention. The primary aim of the study will be to evaluate the hypothesis that AGS, as compared to SGS, results in greater increases over time to four hypothesized psychological mechanisms. The secondary aim will be to evaluate whether post-intervention increases to any among these three mechanisms mediate the relationship between intervention type (AGS vs. SGS) and increases to PA over the course of the intervention.

DETAILED DESCRIPTION:
Interested participants will schedule and complete a phone screen with a researcher to determine eligibility, and if deemed eligible, will complete an initial hour-long baseline assessment with a member of the study team. The baseline assessment will be conducted over video call using the secure, easy-to-use and HIPAA-compliant Zoom service hosted by Drexel University. During the baseline assessment, the assessor will electronically obtain the participant's informed consent to participate in the study, guide the participant on using a mobile phone application to track their daily steps (Google Fit), verbally provide participants with psychoeducational content on safely increasing their physical activity, and administer a psychological task (Implicit Association Test) as well as questionnaires (Demographics; Physical Activity Enjoyment Scale; Treatment Self-Regulation Questionnaire; Self-Efficacy for Exercise Scale). Immediately following the assessment, participants will be randomized to receive one of two possible remote physical activity interventions: adaptive goal-setting (AGS) or static goal-setting (SGS). Randomization will follow a stratified procedure based on age (cutoff point = 45 years), and permuted block randomization will be used within strata to assign individuals to an intervention condition (AGS or SGS). Both interventions will be preceded by a 10-day baseline "run-in" period during which participants will be asked to record their activity but will not receive any daily step goals. In addition, in both interventions, a brief (10-minute) mid-study (3-week) check-in call will be conducted with each participant by a member of the study team to encourage continued compliance with step goals and problem-solve any barriers to increasing physical activity. Participants will also complete a brief survey once each week over the course of the intervention period. At the conclusion of the intervention period, participants will complete several post-intervention questionnaires/tasks and will then be compensated for their participation.

Participants in the adaptive goal-setting condition will begin receiving a new step goal each day over text message (SMS) following the baseline run-in period (starting Week 2). These messages will continue to be delivered each day for the entire duration of the 6-week intervention period (through Week 8), and will contain information about the participant's daily-assigned step goal as well as their number of steps on the previous day in reference to their previous day's goal. Goals will be calculated using a 60th percentile method (consistent with prior research on adaptive goal-setting), such that each day's goal will be set to the 60th percentile value of the last 9 days of available step data for that participant. Goals will be calculated by an algorithm stored on a remote database that automatically extracts user data from the Google Fit cloud server (Google Fitness Store). The database will store daily steps data for each participant, use these data to calculate new daily step goals and transmit them over SMS using a commercial cloud communications platform. The maximum steps goal permitted by the algorithm will be 20,000 steps/day, to ensure that goals remain within an attainable range for most individuals. Participants in the static goal-setting condition will receive the same exact step goal each day (10,000 steps), consistent with prior research, and will receive daily text message updates providing a summary of their previous day's steps and encouraging them to reach their 10,000-step goal for that day.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old
2. Reporting a desire to increase physical activity in order to lose weight, prevent weight gain or improve physical health
3. Possessing a smartphone that can connect to a WiFi (wireless fidelity) network
4. Daily access to a WiFi connection
5. Ability to understand and provide informed consent
6. Proficiency in speaking, reading, and writing English
7. Currently report engaging in insufficient levels of physical activity (<150 minutes/week of moderate-to-vigorous physical activity)

Exclusion Criteria;

1. Present involvement in another physical activity promotion or a behavioral weight loss program
2. Pregnant or planning to become pregnant within the next 6 months (exclude for either)
3. Current BMI <18.5 kg/m^2
4. Diagnosis of a medical condition that could limit the ability to increase physical activity
5. Acute suicide risk (exclude if present in the past 2 weeks or if any attempts were made in past 2 years)
6. Current substance use disorder
7. Current diagnosis of psychosis
8. Current diagnosis of bipolar disorder
9. Currently meet criteria for loss-of-control eating
10. Presence of compensatory behaviors (vomiting, laxatives, diuretics, exercise)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change to Week 3 Expectancy Beliefs about Goals at Week 7 | Measured once weekly from Week 3 through Week 7
  Expectations about one's own ability to achieve physical activity goals will be assessed weekly using a single Likert scale derived from prior research on Expectancy-Values Theories (EVT) of achievement motivation. Responses on the scale will range from 1-5, with higher values representing higher expectations about one's ability to achieve daily activity goals.
Change to Week 3 Affective Appraisals of Goals at Week 7 | Measured once weekly from Week 3 through Week 7
  Appraisals of daily physical activity goals will assessed weekly using a single Likert scale item asking participants to rate their emotional reactions to daily goals on a scale from 1 (Most Negative) to 10 (Most Positive).
Change to Week 3 Perceived Value of Goals at Week 7 | Measured once weekly from Week 3 through Week 7
  Perceived Value of Goals corresponds to the value or importance that an individual attributes to assigned activity goals, and will be assessed weekly using four items derived from Expectancy-Value Theory (EVT) questionnaires (attainment value; interest value; utility value; cost). All items will be measured on a 1-5 Likert scale where higher scores represent higher perceived value, and the mean of all four items will be used to generate an overall Perceived Value score.
Change to Baseline Implicit Attitudes Towards Exercise at Week 8 | Measured at Week 0 (baseline) and Week 8 (post-intervention)
  Implicit attitudes towards exercise will be measured using an Implicit Association Test (IAT) tailored to examine attitudes towards exercise. Image and text stimuli will be closely adapted from prior IAT research in the domain of exercise, with "Exercise" vs. "Not Exercise" serving as the concept dimension and "Pleasant" vs. "Unpleasant" serving as the attribute dimension. A difference score (d-score) will be computed for each participant, with more positive scores indicating more favorable implicit attitudes towards exercise.

SECONDARY OUTCOMES:
Change to Baseline Self-efficacy for Exercise at Week 8 | Measured at Week 0 (baseline) and Week 8 (post-intervention)
  Self-efficacy regarding one's ability to exercise will be examined using the Self-Efficacy for Exercise (SEE) questionnaire. This 9-item questionnaire assesses an individual's confidence in their ability to exercise when faced with a variety of barriers (e.g., fatigue, discomfort, lack of time). Items are rated on a 0-10 scale, with higher scores representing greater self-efficacy about one's ability to exercise. Scores for each item are averaged to compute an overall self-efficacy score.
Change to Baseline Physical Activity Enjoyment at Week 8 | Measured at Week 0 (baseline) and Week 8 (post-intervention)
  Enjoyment of physical activity will be assessed using the Physical Activity Enjoyment Scale (PACES) is an 18-item measure that evaluates enjoyment of various facets of physical activity on a 7-point bipolar Likert scale, with higher scores indicating greater enjoyment of exercise. Scores for each item are averaged to compute an overall physical activity enjoyment score.
Change to Autonomous Motivation to Exercise at Week 8 | Measured at Week 0 (baseline) and Week 8 (post-intervention)
  Autonomous motivation to exercise will be assessed using the Treatment Self-Regulation Questionnaire (TSRQ), which is a 15-item measure examines several facets of motivation to engage in health behaviors as conceptualized by self-determination theory. Responses are rated on a Likert scale (0 = not at all true, 7 = very true) and averaged across items to compute individual subscale scores (autonomous, external, introjected, identified, amotivation). The current study will focus primarily on the Autonomous Motivation subscale, which assesses an individual's intrinsic reasons for engaging in health behaviors.
Change to Baseline Daily Levels of Physical Activity at Week 8 | Measured at Week 0 (baseline) and Week 8 (post-intervention)
  Daily level of physical activity will be measured as the number of steps that a participant records each day using their smartphone pedometers. Daily steps data collected over the full duration intervention phase will be automatically transferred via Google Fit to a remote database where they will be stored and later analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No